CLINICAL TRIAL: NCT02802709
Title: A Placebo-controlled, Double-blind, Randomized Trial of an Intra-articular Device, SB-061, in Symptomatic Osteoarthritis of the Knee
Brief Title: A Trial of SB-061 in Osteoarthritis of the Knee
Acronym: MODIFY-OA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Symic OA Co. (Industry)
Collaborators: Nordic Bioscience Clinical Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TP-1621
Record Dates: First submitted 2016-05-27; First posted 2016-06-16 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis
Keywords: knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB-061 (Experimental): SB-061
  Interventions: Device: SB-061
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Device: SB-061 — delivered via intra-articular injection
  Arms: SB-061
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study evaluates a novel agent, SB-061, for the treatment of osteoarthritis of the knee. Half of the patients will receive the agent via intra-articular injection and half will receive a placebo injection.

DETAILED DESCRIPTION:
The treatment of pain associated with osteoarthritis may include periodic intra-articular injections of corticosteroids or viscosupplements such as hyaluronic acid. SB-061 is anticipated to relieve osteoarthritis pain by reinforcing the cartilage matrix and providing a lubricating coating of the cartilage. Subjects will receive 2 intra-articular injections of either SB-061 or placebo and be followed for 3 months to evaluate pain amelioration. Subjects and Investigators are blinded to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Femorotibial osteoarthritis of the knee
* Radiological OA Kellgren-Lawrence grade 2 or 3
* WOMAC Pain 1 score of the target knee of ≥4 and ≤ 9

Exclusion Criteria:

* Hypersensitivity to medications or to intra-articular injections
* Intra-articular delivery of corticosteroids or hyaluronic acid in the target knee within 6 months of study
* High dose systemic corticosteroid treatment of longer (>14 days) duration w/in 6 months of study
* Major surgery or arthroscopy of the target knee within year prior to study
* Planned surgery in the target knee within the next 3 months
* Concomitant inflammatory disease affecting either knee

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain | Baseline, 3 months
  Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain (A1) scores from baseline to 3 months post treatment will be compared between treatment and control groups.
Incidence of Treatment-Emergent Adverse Events | Through 3 months
  A summary of Treatment-Emergent Adverse Events will be reported

SECONDARY OUTCOMES:
Pain | Baseline, 3 months
  Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) sub-scores scores related to pain from baseline to 3 months post treatment will be compared between treatment and control groups.
Physical function | Baseline, 3 months
  Change in Patient Global Assessement scores from baseline to 3 months post treatment will be compared between treatment and control groups.
Pain | Baseline, 3 months
  Change in Numeric Rating Scale (NRS) of pain from baseline to 3 months post treatment will be compared between treatment and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Bachtell, MD, Study Director — Symic OA Co.
Locations (2):
- Estonia (2):
  - CCBR, Tallinn
  - Medita Kliinik, Tartu

IPD SHARING:
Plan to Share IPD: No